CLINICAL TRIAL: NCT00343616
Title: Investigating Cognitive Function for Patients Participating in the BIG Trial 1-98 in Select Centers
Brief Title: Cognitive Function in Postmenopausal Women With Breast Cancer Receiving Hormone Therapy on Clinical Trial IBCSG-1-98
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000482396; IBCSG-18-98-CFS; IBCSG-1-98-CFS; NOVARTIS-2026703019; EU-20624
Record Dates: First submitted 2006-06-22; First posted 2006-06-23 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Breast Cancer; Cognitive/Functional Effects; Fatigue; Psychosocial Effects of Cancer and Its Treatment
Keywords: cognitive/functional effects; fatigue; psychosocial effects of cancer and its treatment; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Fatigue | interventions — Mental Status and Dementia Tests; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Tamoxifen for 5 years (Experimental): Patients treated with tamoxifen for 5 years after randomization.
  Interventions: Procedure: cognitive assessment; Procedure: fatigue assessment and management; Procedure: psychologic distress; Procedure: quality-of-life assessment
- Letrozole for 5 years (Experimental): Patients treated with letrozole for 5 years after randomization.
  Interventions: Procedure: cognitive assessment; Procedure: fatigue assessment and management; Procedure: psychologic distress; Procedure: quality-of-life assessment
- Tamoxifen 2 years plus letrozole 3 years (Experimental): Patients treated with tamoxifen for 2 years and afterwards with letrozole for 3 years.
  Interventions: Procedure: cognitive assessment; Procedure: fatigue assessment and management; Procedure: psychologic distress; Procedure: quality-of-life assessment
- Letrozole for 2 years plus tamoxifen for 3 years (Experimental): Patients treated with letrozole for 2 years and afterwards with tamoxifen for 3 years.
  Interventions: Procedure: cognitive assessment; Procedure: fatigue assessment and management; Procedure: psychologic distress; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: cognitive assessment — Cognitive function will be assessed using the CogState battery and the Cognitive Failures Questionnaire.
Procedure: fatigue assessment and management — Fatigue will be evaluated using the Brief Fatigue Inventory.
Procedure: psychologic distress — Psychologic distress will be evaluated using the General Health Questionnaire after cognitive testing.
Procedure: quality-of-life assessment — Quality of life will be assessed using global linear analogue self-assessment (LASA) indicators for physical well-being, mood, coping effort (PACIS), perceived social support and subjective health estimation.

SUMMARY:
RATIONALE: Studying cognitive function, such as thinking, attention, concentration, and memory, in postmenopausal women receiving hormone therapy for breast cancer may help improve quality of life and the ability to plan treatment for cancer.

PURPOSE: This phase III trial is studying cognitive function in postmenopausal women with breast cancer receiving hormone therapy on clinical trial IBCSG-1-98.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare cognitive function in postmenopausal women with breast cancer who have received 5 years of adjuvant tamoxifen vs letrozole on protocol IBCSG-1-98.

Secondary

* Compare cognitive function in patients who have received a single hormonal therapy for 5 years vs those who have received that same hormonal therapy for 3 years, having previously received an alternate hormonal therapy for 2 years.
* Compare improvement in cognitive function 1 year after cessation of adjuvant hormonal therapy.
* Compare changes in cognitive function in patients who have received prior adjuvant chemotherapy vs those who have not received adjuvant chemotherapy.
* Assess the relationship between objective and subjective measures of cognitive function, including specific cognitive domains.
* Assess the relationship between cognitive function and psychological distress, fatigue, and quality of life.

OUTLINE: This is a longitudinal, multicenter study.

Patients undergo cognitive function testing and complete self-reported questionnaires regarding cognitive ability, quality of life, fatigue, and psychosocial status during the fifth year of adjuvant hormonal therapy on protocol IBCSG-1-98 and then during the sixth year* (post randomization on protocol IBCSG-1-98) (i.e., after completion of adjuvant hormonal therapy).

NOTE: *Patients who receive extended letrozole, hormone replacement therapy, or other endocrine therapy beyond 5 years do not undergo the 6-year assessment.

PROJECTED ACCRUAL: A total of 148 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Enrolled in protocol IBCSG-1-98

  * Must be in the fifth year of study treatment (i.e., still receiving tamoxifen or letrozole)
* No breast cancer recurrence or second malignancy
* Patients who received 2-4½ years of tamoxifen and have chosen to switch to letrozole to complete 5 years of treatment on protocol IBCSG-1-98 are not eligible
* Hormone receptor status

  * Estrogen receptor- and/or progesterone receptor-positive tumor

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent hormone replacement therapy

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Objective cognitive function as measured by the CogState battery | 6 years after randomization

SECONDARY OUTCOMES:
Subjective cognitive function as measured by the Cognitive Failures Questionnaire (CFQ) | 6 years after randomization
Psychological distress as measured by the General Health Questionnaire (GHQ) | 6 years after randomization
Fatigue as measured by the Brief Fatigue Inventory (BFI) | 6 years after randomization
Quality of life as measured by the IBCSG QL Core Form | 6 years after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Kelly-Anne Phillips, Study Chair — Peter MacCallum Cancer Centre, Australia; Juerg Bernhard, PhD, Study Chair — ETOP IBCSG Partners Foundation
Locations (12):
- Australia (4):
  - Institute of Oncology at Prince of Wales Hospital, Randwick, New South Wales
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St. Vincent's Hospital - Melbourne, Fitzroy, Victoria
  - Cabrini Hospital, Malvern, Victoria
- Institut Jules Bordet, Brussels, Belgium
- European Institute of Oncology, Milan, Italy
- Auckland City Hospital, Auckland, New Zealand
- Switzerland (4):
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona
  - International Breast Cancer Study Group, Bern
  - Kantonsspital - St. Gallen, Sankt Gallen
- Ninewells Hospital, Dundee, Scotland, United Kingdom